CLINICAL TRIAL: NCT00880750
Title: A Phase I Pharmacodynamic Equivalence Study Comparing Urinary Phosphate Excretion and Plasma Lanthanum Pharmacokinetics for a Lanthanum Carbonate Granule Formulation and Chewable Tablets Administered to Healthy Adult Subjects
Brief Title: Pharmacodynamic Study of Two Lanthanum Carbonate Formulations in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD405-127
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: End Stage Renal Disease
Keywords: End stage Renal disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lanthanum carbonate granules (Experimental): Lanthanum carbonate granulated formulation crossover to chewable tablet formulation
  Interventions: Drug: Lanthanum carbonate Granule Formulation
- Lanthanum carbonate chewable tablets (Fosrenol) (Experimental): Lanthanum carbonate chewable table formulation crossover to granulated formulation
  Interventions: Drug: Lanthanum carbonate Chewable Tablets (Fosrenol)

INTERVENTIONS:
Drug: Lanthanum carbonate Granule Formulation — 3x's per day for 3 days, 1 dose in the am for day 4. (A single dose equals 1000mg of lanthanum carbonate granule formulation. Dose is administered immediately after each meal.)
  Arms: Lanthanum carbonate granules
Drug: Lanthanum carbonate Chewable Tablets (Fosrenol) — 3x's per day for 3 days, 1 dose on day 4. (A single dose equals a 1000mg tablet of lanthanum carbonate. Dose is administered immediately after each meal.)
  Other Names: Fosrenol
  Arms: Lanthanum carbonate chewable tablets (Fosrenol)

SUMMARY:
This study is being conducted to assess any potential differences in the absorption and excretion between two lanthanum carbonate formulations. This study is also being done to assess the safety and tolerability of the two lanthanum carbonate formulations.

ELIGIBILITY:
Inclusion Criteria

* Ability to provide informed consent to participate in the study.
* Healthy volunteers, age 18-55 inclusive.
* Subject must be willing to comply with applicable contraceptive requirements of the protocol
* Female subjects must have a negative pregnancy test
* Ability to chew and or swallow doses of the investigational products as prescribed in the protocol.
* Ability to fully comply with all study procedures and restrictions, including consumption of all food provided while a resident in the CRC.

Exclusion Criteria

* Current or relevant previous history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or study procedures.
* Clinically significant abnormal serum phosphate levels, outside of normal limits.
* Current use of any medication with the exception of hormonal replacement therapy or hormonal contraceptives within 7 days of first dose of investigational product.
* A known history of lactose intolerance or allergy to milk or other foods.
* Clinically significant or multiple allergies as determined by an Investigator.
* History of alcohol or other substance abuse within the last 6 months.
* A positive screen for alcohol or drugs of abuse.
* Male subjects who consume more than 21 units of alcohol per week or three units per day. Female subjects who consume more than 14 units of alcohol per week or two units per day.
* A positive human immunodeficiency virus (HIV) antibody screen, Hepatitis B surface antigen (HBsAg) or Hepatitis C virus (HCV) antibody screen.
* Female subjects who are pregnant (positive pregnancy test), lactating, or less than 90 days post-partum.
* Subjects that have previously been randomized in this study.
* Use of tobacco in any form or other nicotine-containing products in any form. Ex-users must report that they have stopped using tobacco for at least 60 days prior to receiving the first dose of investigational product.
* Routine consumption of more than two units of caffeine per day or subjects who experience caffeine withdrawal headaches.
* Donation of blood or blood products within 60 days prior to receiving the first dose of investigational product.
* Plasma donation within 28 days prior to the first dose of the investigational product.
* Use of another investigational product within 30 days prior to receiving the first dose of investigational product or active enrolment in another drug or vaccine clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-01-28 (Actual); Primary Completion 2009-06-22 (Actual); Study Completion 2009-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- West Coast Clinical Trials, LLC, Cypress, California, United States

REFERENCES:
- [Result] Pierce D, Hossack S, Robinson A, Zhang P, Martin P. Assessment of pharmacodynamic equivalence and tolerability of lanthanum carbonate oral powder and tablet formulations: a single-center, randomized, open-label, 2-period crossover study in healthy subjects. Clin Ther. 2012 Jun;34(6):1290-1300.e2. doi: 10.1016/j.clinthera.2012.05.003. Epub 2012 May 31. PMID 22657252
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Lanthanum Carbonate Granules First: Granule formulation first at 1000 mg three times a day for 3 days and a single 1000 mg dose after breakfast on Day 4, a washout period, then chewable tablet formulation at 1000 mg three times a day for 3 days and a single 1000 mg dose after breakfast on Day 4.
- Lanthanum Carbonate Chewable Tablet First: Chewable tablet formulation first at 1000 mg three times a day for 3 days and a single 1000 mg dose after breakfast on Day 4, a washout period, then granule formulation at 1000 mg three times a day for 3 days and a single 1000 mg dose after breakfast on Day 4.
Period: First Intervention
Arm/Group | Lanthanum Carbonate Granules First | Lanthanum Carbonate Chewable Tablet First
Started | 39 | 33
Completed | 30 | 32
Not Completed | 9 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Unable to collect urine | 4 | 0
Not completed — Non-compliance with meals | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Washout Period
Arm/Group | Lanthanum Carbonate Granules First | Lanthanum Carbonate Chewable Tablet First
Started | 30 | 32
Completed | 30 | 32
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Lanthanum Carbonate Granules First | Lanthanum Carbonate Chewable Tablet First
Started | 30 | 32
Completed | 26 | 30
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Unable to collect urine | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanthanum Carbonate Granules First | Lanthanum Carbonate Chewable Tablet First | Total
Number analyzed (Participants) | 39 | 33 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 33 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (8.70) | 31.3 (7.83) | 31.4 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 28 | 24 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 33 | 72

OUTCOME MEASURES:

1. Primary Outcome: Urinary Phosphate Excretion 3-Day Average
Time Frame: Continuous collection over 3 days
Population: Pharmacodynamic Set (PD) includes all subjects who completed all urine collections and consumed at least 95% of food in all treatment periods. Subjects who vomited from days -2 to 4 of any treatment period were excluded from the set.
Measure: Least Squares Mean (Standard Error); unit: mmol
Groups:
- Lanthanum Carbonate Granules: Granule formulation at 1000 mg three times a day for 3 days and a single 1000 mg dose after breakfast on Day 4
- Lanthanum Carbonate Chewable Tablet: Chewable tablet formulation at 1000 mg three times a day for 3 days and a single 1000 mg dose after breakfast on Day 4
Arm/Group | Lanthanum Carbonate Granules | Lanthanum Carbonate Chewable Tablet
Number analyzed (Participants) | 49 | 49
mmol | 16.01 (0.485) | 17.35 (0.484)
Statistical Analysis 1: Comparison: Lanthanum Carbonate Granules vs Lanthanum Carbonate Chewable Tablet; Test type: Non-Inferiority or Equivalence — A standard 90% confidence interval (CI) was constructed for the difference in least square means of the primary pharmacodynamic (PD) variable between the granules formulation and the reference chewable tablet formulation. A critical reference representing +/- 20% of the reference chewable tablet formulation least squares mean was constructed. PD equivalence was to be claimed if the 90% CI was completely contained within the critical reference range of (-3.47, 3.47); Mixed Models Analysis; Mean Difference (Final Values) = -1.35, 90% CI 2-sided [-2.18 to -0.51]

2. Secondary Outcome: Urinary Phosphate Excretion on Day 4
Time Frame: Continuous collection on Day 4
Population: PD set
Measure: Least Squares Mean (Standard Error); unit: mmol
Arm/Group | Lanthanum Carbonate Granules | Lanthanum Carbonate Chewable Tablet
Number analyzed (Participants) | 49 | 49
mmol | 15.03 (0.569) | 17.01 (0.569)
Statistical Analysis 1: Comparison: Lanthanum Carbonate Granules vs Lanthanum Carbonate Chewable Tablet; Test type: Non-Inferiority or Equivalence — A standard 90% confidence interval (CI) was constructed for the difference in least square means of the primary pharmacodynamic (PD) variable between the granules formulation and the reference chewable tablet formulation. A critical reference representing +/- 20% of the reference chewable tablet formulation least squares mean was constructed. PD equivalence was to be claimed if the 90% CI was completely contained within the critical reference range of (-3.40, 3.40); Mixed Models Analysis; Mean Difference (Final Values) = -1.98, 90% CI 2-sided [-3.17 to -0.80]

3. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of Lanthanum Carbonate
Time Frame: 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose on Day 4
Population: Pharmacokinetic set (PK) includes all subjects who had sufficient post-dose blood samples taken to estimate Cmax and AUC 0-48 hours after dosing on Day 4 in all treatment periods. Subjects who vomited between dosing and 10 hours post-dose on Day 4 of any treatment period were excluded from the PK set.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Lanthanum Carbonate Granules | Lanthanum Carbonate Chewable Tablet
Number analyzed (Participants) | 62 | 58
ng*h/ml | 14.2 (6.02) | 10.3 (3.50)
Statistical Analysis 1: Comparison: Lanthanum Carbonate Granules vs Lanthanum Carbonate Chewable Tablet; The LS means and associated SEs for granules and tablets as well as the difference between granules and tablets were determined. From the LS mean and SE of the difference, a 90% CI was constructed for the difference of the logs of granules and tablets. An exponential transformation was applied to the lower and upper limits of the CI. This created a point estimate and 90% CI for the ratio of LS means for granules to tablets; Test type: Superiority or Other; Mixed Models Analysis; After application of the log transformation AUC 0-48 was analysed using a mixed effect linear model; Ratio of geometric LS means = 1.34, 90% CI [1.26 to 1.42]

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lanthanum Carbonate
Time Frame: 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose on Day 4
Population: PK set
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lanthanum Carbonate Granules | Lanthanum Carbonate Chewable Tablet
Number analyzed (Participants) | 64 | 58
ng/ml | 0.638 (0.241) | 0.504 (0.181)
Statistical Analysis 1: Comparison: Lanthanum Carbonate Granules vs Lanthanum Carbonate Chewable Tablet; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; After application of the log transformation Cmax was analysed using a mixed effect linear model; Ratio of geometric LS means = 1.26, 90% CI [1.20 to 1.33]

5. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Lanthanum Carbonate
Time Frame: 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose on Day 4
Population: PK set
Measure: Median (Full Range); unit: hours
Arm/Group | Lanthanum Carbonate Granules | Lanthanum Carbonate Chewable Tablet
Number analyzed (Participants) | 64 | 58
hours | 4.00 (0.0) [0 to 6.00] | 4.00 (0.0) [0 to 8.00]
Statistical Analysis 1: Comparison: Lanthanum Carbonate Granules vs Lanthanum Carbonate Chewable Tablet; Test type: Superiority or Other; Wilcoxon (Hodges-Lehmann); The median difference and 90% CI for the median difference was then calculated based on Hodges-Lehmann estimate for Wilcoxon's Signed Rank test; Median Difference (Final Values) = 0.01, 90% CI [0.00 to 0.50]

ADVERSE EVENTS:
Description: Safety set (SS) consists of subjects who received at least 1 dose of the investigational medicinal product and had at least 1 post-dose safety assessment.
Arm/Group | Lanthanum Carbonate Granules | Lanthanum Carbonate Chewable Tablet
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/61
Other Adverse Events (participants affected / at risk) | 9/71 | 6/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanthanum Carbonate Granules (N=71) | Lanthanum Carbonate Chewable Tablet (N=61)
Nausea (Gastrointestinal disorders) | 6 (7) | 3 (3)
Headache (Nervous system disorders) | 4 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.